CLINICAL TRIAL: NCT00497341
Title: Randomised And Double Blind Study To Evaluate The Best Moment To Infuse The Prophylactic Antibiotic In Knee Arthroplasty Performed Under Ischemia
Brief Title: Antibiotic Prophylaxis in Total Knee Prosthesis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Alex Soriano, Consultant of infectious diseases, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: PTR2007
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Infection
Keywords: infection after total knee arthroplasty
MeSH Terms: conditions — Infections | interventions — Cefuroxime

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): antibiotic is given before tourniquet inflation and before tourniquet release
  Interventions: Drug: cefuroxime
- 2 (Placebo Comparator): antibiotic is given before tourniquet inflation
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: cefuroxime — cefuroxime is administered at a dosage of 1.5 g before tourniquet inflation and release in experimental arm and only before tourniquet inflation in control arm
  Arms: 1
Drug: placebo — cefuroxime 1.5 g IV before tourniquet inflation + placebo before tourniquet release + cefuroxime 1.5 g IV 6 h after surgery
  Arms: 2

SUMMARY:
Knee prosthesis infection is a severe complication. The use of a tourniquet during surgery impairs the efficacy of the antibiotic prophylaxis. We hypothesize that the antibiotic administration before tourniquet release decrease the infection rate. Methods: patients who undergo a total knee arthroplasty will be randomized to receive one of the following regimens of antibiotic prophylaxis:Standard: cefuroxime 1.5 g i.v. 10 min before tourniquet + placebo 10 min before tourniquet release + cefuroxime 1'5 g i.v. 6h after closing surgical wound.Experimental: cefuroxime 1.5 g i.v. 10 min before tourniquet + cefuroxime 1.5 g i.v. 10 min before tourniquet release + cefuroxime 1'5 g i.v. 6h after closing surgical wound.

DETAILED DESCRIPTION:
Objective: when surgery is performed under ischemia, the ideal timing for the administration of antibiotic prophylaxis has not been well defined. Currently, antibiotics are given 10 minutes before ischemia and the infection rate is about 3-5%. In 2005 we performed a study where the efficacy of the standard prophylaxis was compared with a new regimen that consisted in administering the antibiotic 10 min. before tourniquet release. The results were positive although the difference was not statistically significant. In the present study we are proposing a new protocol where the antibiotic is given 10 min. before the inflation of tourniquet and 10 min. before its release. Methodology: all patients who undergo a total knee arthroplasty will be randomized to receive one of the following regimens of antibiotic prophylaxis:Standard: cefuroxime 1.5 g i.v. 10 min before tourniquet + placebo 10 min before tourniquet release + cefuroxime 1'5 g i.v. 6h after closing surgical wound.Experimental: cefuroxime 1.5 g i.v. 10 min before tourniquet + cefuroxime 1.5 g i.v. 10 min before tourniquet release + cefuroxime 1'5 g i.v. 6h after closing surgical wound.The infection rate with standard regimen is 3.4%. We believe that the new regimen will decrease the rate of infection to 1%. To demonstrate differences between both arms, it will be necessary to include 666 patients per arm.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing knee arthroplasty

Exclusion Criteria:

* patients allergic to penicillin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1332 (Actual)
Dates: Start 2008-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
infection rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alex Soriano, MD, Principal Investigator — Hospital Clínical
Locations (1):
- Hospital Clínic, Barcelona, Catalonia, Spain